CLINICAL TRIAL: NCT06599255
Title: One-Puncture Versus Multipoint Technique of Rectus Sheath Block With Transverse Abdominis Plane Block for Analgesia After Laparoscopic Cholecystectomy
Brief Title: One-Puncture Versus Multipoint Technique of Rectus Sheath Block With Transverse Abdominis Plane Block
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Mohamed Medhat, assistant professor of anesthesia and surgical intensive care (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB#568/27-AUG-2024
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- one puncture (Active Comparator): one-puncture technique of RSB combined with TAPB.
  Interventions: Procedure: US-guided RSB and TAPB by one-puncture technique.
- Multipoint (Active Comparator): multipoint technique of RSB combined with TAPB.
  Interventions: Procedure: multipont
- control (No Intervention): nalbuphine (2 mg/kg) and normal saline to a total volume of 150 mL, with a background infusion rate of 2 mL/h, a bolus dose of 2 mL, a lockout interval of 15 min, and a maximum limit of 10 mL within 1 h.

INTERVENTIONS:
Procedure: US-guided RSB and TAPB by one-puncture technique. — The probe will be positioned transversely in the midline of the abdomen, between the xiphoid process and the umbilicus, revealing the linea alba. It was then moved outward along the costal margin, demonstrating the rectus abdominis overlapping the transverse abdominis. A 22-gauge, 120-mm ultrasound-visible block needle will be inserted from the inner side . Under direct vision, we will reach the posterior rectus abdominis sheath and pierced the anterior layer of the posterior sheath. Saline was injected to adjust its position. After that, 15 mL of 0.25% bupivacaine will be administered (aspiration was performed for every 5 mL injection), and we will observe the local anesthetic spreading inward . Then, the needle will break through the posterior layer of the tendon, and saline will be injected to confirm the needle's placement in the transversus abdominis plane. After confirming the tip placement, 15 mL of 0.25% bupivacaine will be slowly injected. The needle tip will be advanced al
  Arms: one puncture
Procedure: multipont — , the probe will be moved outward along the costal margin until the external oblique muscle, internal oblique muscle, and transverse abdominis muscle will be visible [9]. The needle will be inserted in-plane until the tip was positioned in the plane between the internal oblique muscle and the transverse abdominis muscle. Then, 15 mL of 0.25% bupivacaine will be injected . The contralateral nerve block will be performed using the same method and volume of anesthetic solution.
  For the RSB, the same technique will be done as one puncture technique. Then, 15 mL of 0.25% bupivacaine will be injected . The contralateral nerve block will be performed using the same method and volume of anesthetic solution.
  Arms: Multipoint

SUMMARY:
the purpose of this study is to compare of better postoperative analgesia following laparoscopic cholecystectomy using either one puncture rectus sheath block with transverse abdominis plane block or multipoint technique

DETAILED DESCRIPTION:
after being informed about the study and potential risks. All patients giving written consent will be randomized by double blind manner into 3 groups each one containing 34In the One puncture "O" group (n= 34): The patient will receive one-puncture technique of RSB combined with TAPB.

In the Multipoint "M " group (n= 34): The patient will receive multipoint technique of RSB combined with TAPB.

In the Control "C " group (n=34 ): The patient will receive patient controlled analgesia&;PCA&

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old.
* Sex: both sexes.
* Physical status: ASA I to III.
* Body mass index (BMI): 18- 30 kg/m2.
* Type of operations: elective laparoscopic cholecystectomy.
* Written informed consent from the patient.

Exclusion Criteria:

* Known hypersensitivity to lidocaine or bupivacaine.
* Opioid-dependent patients.
* Coagulation disorders or taking drugs affect surgical hemostasis.
* Patients with pre-existing neurological deficits.
* Uncooperative patient or with altered mental status.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The total postoperative opioid consumption in the first 24 hours. | 24 hours postoperative
  opioid consumption

SECONDARY OUTCOMES:
The block performance time | up to 5 minutes
  the time from the placement of the ultrasound probe on the patient's skin to the end of the local anesthetic injection
Onset of sensory block | up to 30 minutes
  the time from the end of the injection of local anesthetic (bupivacaine) to the loss of pinprick sensation using a sterile 25-G needle in the operation field.
The Numerical Pain Rating Scale | 24 hours postoperative
  A ten-centimeter Numerical Pain Rating Scale (0 - no pain and 10 - worst pain)
Patient satisfaction | 24 hour postoperative
  The patient satisfactionwill be assessed using the 7-point Likert-like verbal rating scale The patientwill be asked to express his satisfaction
  1. extremely dissatisfied.
  2. Dissatisfied.
  3. somewhat dissatisfied.
  4. unsatisfied.
  5. somewhat satisfied.
  6. Satisfied.
  7. extremely satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine,Zagazig University, Zagazig, Elsharkia,, Egypt,, Egypt

IPD SHARING:
Plan to Share IPD: No